CLINICAL TRIAL: NCT05833503
Title: Efficacy Study of Two Types of Intervention for People in Couple Who Have Difficulties With Their Gambling Habits or Alcohol/Drug Use
Brief Title: Integrative Couple Treatment for Gambling/Substance Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Collaborators: Université du Québec a Montréal (Other); Université de Sherbrooke (Other); Laval University (Other); Université de Montréal (Other)
Responsible Party: Principal Investigator, Joël Tremblay, PhD. Professor to department of psychoeducation, Université du Québec à Trois-Rivières
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FRQSC-2022-0JUL-307826
Record Dates: First submitted 2023-02-10; First posted 2023-04-27 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Gambling Disorder; Substance Use Disorders
Keywords: Gambling Disorder; Substance use Disorder; Couple-based intervention; Marital relationship
MeSH Terms: conditions — Gambling; Substance-Related Disorders | interventions — Couples Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either Integrative Couple Therapy for Addiction (ICT-A, experimental group) or the usual individual treatment (control group).
Masking Description: These are two behavioral treatments.It is therefore impossible to mask the allocation of participants to either treatment, for both participants and clinicians.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrative Couple Treatment for Addiction (ICT-A) (Experimental): Inspired by the "Alcohol Behavior Couple Therapy" from Epstein & McCrady, the ICT-A will be offered over 12 to 16 sessions of 90 minutes. Typically, approximately the first half of each session is dedicated to GD/SUD problems,in a predominantly cognitive behavioral model. In the second part of each session, the clinician will help the couple to improve their communication,to reduce the reinforcements (non-voluntary) of the behaviors of GD/SUD and to increase marital pleasure situations incompatible with the use of GD/SUD.Particular attention will also be paid to feelings of betrayal and interpersonal attacks to restore trust. Plus,they will received a sefl-care guide.
  Interventions: Behavioral: Integrative Couple Treatment for Addiction (ICT-A)
- Individual treatment as usually offered (Active Comparator): The usual treatment control group will receive individual treatment as already offered by the specialized centres in addiction.
  For the person with GD/SUD, this treatment consists of 12 to 16 individual cognitive-behavioral sessions of 60 minutes. In general, the intervention aims to secure financial assets, awareness of erroneous thoughts and improvement of alternative skills to gambling in order to meet the normal demands of psychic and relational life. People undergoing this intervention will receive a self-care guide.
  As for the partners randomized in this intervention, they will receive the services that are usually offered to members of the entourage of a person with GD/SUD. In groups or individually, these services are generally aimed at improving the partner's well-being and relationship with their spouse, which includes information about GD/SUD and the recovery process.
  Interventions: Behavioral: Treatment individual as usually offered

INTERVENTIONS:
Behavioral: Integrative Couple Treatment for Addiction (ICT-A) — Couple-based intervention called Integrative Couple Treatment for Addiction (ICT-A).
  Other Names: Couple therapy
  Arms: Integrative Couple Treatment for Addiction (ICT-A)
Behavioral: Treatment individual as usually offered — Individual-based treatment as usually offer by the specialized centres in addiction.
  Other Names: Treatment as usual (TAU)
  Arms: Individual treatment as usually offered

SUMMARY:
The aim of the study is to compare couple-based treatment to individual treatment (treatment as usual) for addiction (gambling or substance use disorder).

DETAILED DESCRIPTION:
Background:Couple-based intervention is one of the clinical innovations to increase access, retention and effectiveness of treatment in the field of addiction.Couple-based intervention for the treatment of problems related to gambling or substance use disorder (GD/SUD) is more effective than no treatment and the subjective experience of the members of the couple illustrates important clinical gains (better understanding addiction, resolve conflicts, etc.). A study conducted by the research team revealed a better effectiveness of couple-based treatment for GD than the individual treatment usually offered. Despite these positive results, this study highlighted a need to improve the couple intervention model (Integrative Couple Treatment for Pathological Gambling- ICT-PG). First of all, it did not allow to reach people having a SUD. Previous studies conducted by the research team also illustrated the need for more clinical work on serious relationship injuries caused by gambling. The investigators also accentuated their work on the strategies used by the partners and having an impact on the gambler's gambling behaviors.

Goal : Evaluate the effectiveness of a couple-based treatment (Integrative Couple Therapy for Addiction ICT-A; experimental group) compared to the individual treatment usually offer (control group) for people with GD/SUD.

Method/Design : A sample of at least 100 couples will be randomized to either ICT-A (experimental group) or the usual individual treatment (control group). The couple treatment called Integrative Couple Therapy for Addiction (ICT-A) is inspired by the "Alcohol Behavior Couple Therapy" from Epstein and McCrady, to which the team added diverse components to adjust to gamblers. During the sessions, the focus is on a) reducing/stopping gambling or substance use behaviors, b) helping the partner to stop behaviors facilitating gambling habits or substance use and rise the frequency of behaviors incompatible with gambling habits or substance use c) improve marital components (communication, sharing positive moments, negotiation, mutual support).The control group receives individual treatment as already offered by the specialized centers in addiction. All participants are recruited in Specialized Addiction Treatment Centers in Quebec Province, Canada. Repeated measures will be conducted at admission, 6, 12 and 18 months post-admission on the addiction's severity (primary outcome), on various couples' dimensions (secondary outcome) and various indicators of personal well-being (secondary outcome).In order to compare the effectiveness of the two treatment modalities, a series of regression analyzes will be carried out taking into account the correlation between the observations for the same individual and measurements repeated over time (linear mixed models; PROC MIXED of SAS).

ELIGIBILITY:
Inclusion Criteria:

* The Gambler may have a gambling or substance use problem at the beginning of treatment AND is accepted for treatment by addiction rehabilitation centers (CRDs).
* The Gambler has engaged in gambling or substance use behaviors in the past three months (Time Line Follow-Back).
* The Partner may or may not engage in gambling, consume alcohol or other substances of abuse.
* Living in couple for at least six months OR report being in a significant relationship for at least two years.
* Neither member of the couple presents a mental health problem that could hinder their ability to participate in the therapeutic process.

Exclusion Criteria:

* The Gambler has been completely abstinent from any gambling or substance use problem for the past three months.
* The Gambler received treatment for gambling disorder or substance abuse disorder during the last six months (excluding Gamblers Anonymous, Alcoholics Anonymous or Narcotics Anonymous).
* Low level of marital commitment between the couple in the past 2 weeks indicating a high risk of short-term separation (Marital Status Inventory, score ≥9)
* Presence of serious acts of violence committed within the past year endangering the safety or life of one of the spouses (Modified Conflict Tactics Scales: Answer YES to any question from Q27-33) OR use of services for victims of domestic violence in the past year.
* Presence of an active mental health disorder in either partner hindering therapeutic participation, such as a psychotic disorder OR a suicide attempt in the last 30 days (Psychological Scale of the Addiction Severity Index) OR severe borderline personality disorder (BSL-23 ≥2.8) OR excessively extreme antisocial behaviors (Conduct Disorder Scale from the GAIN ≥ 9).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in Self-reports of alcohol, substance use and gambling with the Time-Line Follow-Back (TLFB) in the last 90 days-Gamblers | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  The TLFB evaluates the frequency and quantity of substance consumed (alcohol, cannabis, other drugs) and gambling behaviours in the last 90 days, based on the personal definition of each user (none, low, moderate, high).
Change in Canadian Problem Gambling Severity Index (PGSI)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  The Canadian Problem Gambling Index (CPGI) is a 9-item measure with a 4-point Likert-type scale (0 = Never, 3 = Almost always). It asks questions about the gambler's habits from four categories:
  Gambling involvement; Problem gambling behaviour; Adverse Consequences; Correlates of problem gambling.
  Scores for the nine items are summed, and the results are interpreted as follows: 0 = non-problem ; 1-4 = low risk; 5-7 = moderate risk; 8 and + (maximum 27) = probable pathological player.
Change in Alcohol, Smoking and Substance involvement and Screening Test (ASSIST) of the World Health Organization (WHO)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  This 8-item tool is developed by a group of the World Health Organization (WHO) specialized in addiction. It detects the use of different substances from the gambler and proposes a threshold above which reported consumption behaviors are problematic (low risk: 0-3 for drug use and 0-10 for alcohol use, moderate risk: between 4-26 for drug use and between 11-26 for alcohol use, high risk 27 and more for alcohol and drug use).
Change in Negative Gambling/Using Consequences-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  This short questionnaire of 7 items assesses to what extent the respondent considers his gambling/using habits in the last 3 months have harmed various aspects of his life (financial, living conditions, marital, physical health, professional life, social, legal and family).
  Participants are asked to respond on a scale where "0" corresponds to "not at all" or "never", while "10" corresponds to "extremely" or "always".
  To compute a total score, all item' score are summed. The total score ranges from 0 to 70.The higher the score, the more it indicates that the person is experiencing negative impacts due to their GD/SUD.
Change in Negative Gambling/Using Consequences-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Partners
  This short questionnaire of 7 items assesses to what extent the respondent considers that his partner's gambling/using habits have harmed various aspects of his life in the last 3 months (financial, living conditions, marital, physical health, professional life, social, legal and family).
  Participants are asked to respond on a scale where "0" corresponds to "not at all" or "never", while "10" corresponds to "extremely" or "always".
  To compute a total score, all item' score are summed. The total score ranges from 0 to 70. Higher the score is, more it's indicate that the respondent is experiencing negative impacts because of his partner's gambling habits.
Change in Severity of dependance scale (SDS)-Gamblers | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  This brief questionnaire is designed to measure the severity of a person's addiction. The tool includes 5 items concerning the psychological dimensions of addiction (loss of control, concern about use or gambling behaviors).
  Each question is scored either 0 (Never or almost never),1(Sometimes), 2 (Often), or 3 (Always).
  A total score is calculated by summing the responses to all five questions. The minimum total score possible is 0, and the maximum total score possible is 15 (i.e. total score range: 0-15). A higher total score indicates a higher level of dependence.
Change in Craving Experience Questionnaire (CEQ)-Gamblers | in the last seven days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  The CEQ was developed based on intrusion theory, which conceives of craving as a cognitive-emotional phenomenon that begins with an intrusive and generally spontaneous thought (triggered by external or internal cues) followed by a cognitive process involving the construction of multi-sensory images. The CEQ-forces cravings consists of 10 items assessing craving intensity, images, and thought intrusion. The 4 items covering imagery, scent, taste and mouth/throat sensation have been adapted into three items to better reflect the experience of craving with gambling.
  The CEQ is a 10-items questionnaire that measures the intensity craving (i.e. the irrepressible urge to consume a substance) in the last 7 days. Each item is rated from 0 (Not at all) to 10 (Extremely). Total scores summarise strength of craving, which can range between 0 and 100. The higher the score, the more the craving felt by the participant is considered intense.
Change in Readiness to Change Questionnaire (RCQ)-Gamblers | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  The RCQ is a 12-item instrument used for identifying the "stage of change" of someone having an addiction problem, which are : precontemplation (PC), contemplation (C) and action (A).
  Questions assess the degree of motivation to change substance use and/or gambling habits. The respondent answers with -2 (Strongly disagree), -1 (Disagree), 0 (Unsure), +1 (Agree), +2 (Strongly Agree). The item score for each scale (PC, C and A) is summed, meaning the total score should be within the range -8 to +8. The scale with the highest score is the one that determines the stage of motivation to change.
Change in Readiness Ruler tool-Gambler | in the last seven days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  The instrument has two items, one to estimate how important people with problematic use feel it is to change their behaviors, and another to estimate how capable they feel they are of changing their behaviors, reflecting their sense of competence in changing their behavior or their perceived ability to change.Responses are distributed along a continuum from 0 to 10 where "0" represents "not at all," "5" means "moderately" and "10" represents "extremely."
  Higher the score is for each scale, respectively, the higher the level of importance and the level of confidence about making this change.
Change in Global Improvement Rate-Gambler | in the last six months of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  This scale (of one question only) is used to document the perceived improvement in terms of difficulties in controlling one's gambling and substance use behaviors according to the treatment received. On a 7-point Likert scale (1 = very great degradation; 4 = no change; 7 = very great improvement), the individual evaluates the extent to which he has changed their gambling and substance use compared to prior the treatment.
  The closer the score is to 7, the more progress the person feels he or she has made, while a score close to 4 indicates no change and a score close to 1 indicates that the situation has worsened (max=7, min=0).
Change in Global Improvement Rate-Partner | in the last six months of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  This scale (with a single question) is used to document the improvement perceived by the partner about his gambler spouse in terms of difficulties in controlling his gambling and consumption behaviors according to the treatment received. On a 7-point Likert scale (1 = very great degradation; 4 = no change; 7 = very great improvement). The individual assesses the extent to which his or her partner has changed his or her gambling and substance use patterns from before treatment.
  The closer the score is to 7, the more the person feels that his or her spouse has made progress, while a score close to 4 indicates no change and a score close to 1 that the situation has deteriorated (max=7, min=0).
Change in Inventory of Erroneous Beliefs Related to Gambling ("Inventaire Des Croyances liées Aux Jeux" - ICROLJ)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  This questionnaire measures people's beliefs about gambling. The ICROLJ has 30 items and uses a 4-point Likert-type scale ranging from "Strongly disagree" = 0 to "Strongly agree"=4. To compute a total score, all item' score are summed. The total score ranges from 0 to 120.Higher the score is, more it indicates the presence of erroneous beliefs.
Change in Inventory of Erroneous Beliefs Related to Gambling ("Inventaire Des Croyances liées Aux Jeux" - ICROLJ)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Partners
  This questionnaire measures people's beliefs about gambling. The ICROLJ has 30 items and uses a 4-point Likert-type scale ranging from "Strongly disagree" = 0 to "Strongly agree"=4.
  To compute a total score, all item' score are summed. The total score ranges from 0 to 120. Higher the score is, more it indicates the presence of erroneous beliefs.
Change in integrative evaluation specialized in addiction (évaluation intégrative spécialisée en dépendance)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  This questionnaire measures different dimensions of the addiction problem (consequence, psychic invasion, preoccupation, loss of control, craving, withdrawal, unpleasant emotional motivation). Generally composed of 18 items, we removed the items that were already in the questionnaire on consequences, for a total of 13 items scored on a scale from 0 to 10 (0= not at all, 10=extremely).
  To compute a total score, all item' score are summed. The total score ranges from 0 to 130. The higher the score, the more severe the disorder.

SECONDARY OUTCOMES:
Change in Affective Reserve-Gambler | in the last seven days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  This 2-item questionnaire measures one's emotional reserve and/or affective resources in a relationship. The following questions : 1) " Over the past week, how much have you done to please your partner? " and 2) " Over the past week, what was your level of affective reserve towards your partner? " are answered on a 11-point scale ranging from 0 (never) to 10 (extremely). The higher the score, the more it indicates that the emotional reserve is high (max=20, min=0).
Change in Affective Reserve-Partner | in the last seven days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Partners
  This 2-item questionnaire measures one's emotional reserve and/or affective resources in a relationship. The following questions : 1) " Over the past week, how much have you done to please your partner? " and 2) " Over the past week, what was your level of affective reserve towards your partner? " are answered on a 11-point scale ranging from 0 (never) to 10 (extremely). The higher the score, the more it indicates that the emotional reserve is high (max=20, min=0).
Change in Conflict Tactics Scale-2_Psychological Violence Issued by the Spouse-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  The psychological violence suffered is a subscale of the CTS-2 questionnaire which aims to assess the manifestations of psychological violence committed against the Gambler in the last 3 months. It is made up of 14 items that are rated on a 7-point Likert scale (never happened = 0, 1 time = 1, 2 times = 2, 3 to 5 times = 3, 6 to 10 times = 4, 11 to 20 = 5, more than 20 times = 6). To compute a total score, all item' score are summed. The total score ranges from 0 to 84. The higher it is, more it indicates that the respondent has suffered episodes of psychological violence.
Change in Conflict Tactics Scale-2_Psychological Violence Issued by the Spouse-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  The psychological violence suffered is a subscale of the CTS-2 questionnaire which aims to assess the manifestations of psychological violence committed against the Gambler in the last 3 months. It is made up of 14 items that are rated on a 7-point Likert scale (never happened = 0, 1 time = 1, 2 times = 2, 3 to 5 times = 3, 6 to 10 times = 4, 11 to 20 = 5, more than 20 times = 6). To compute a total score, all item' score are summed. The total score ranges from 0 to 84. The higher it is, more it indicates that the respondent has suffered episodes of psychological violence.
Change in Marital Status Inventory (MSI)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  The MSI is used to measure marital stability in a couple. It comprises a series of 14 items (with inverted items) in a "true" or "false" format thus aiming to assess the risk of separation in this couple (e.g., I very often have ideas of divorce, until once a week or more). Marital distress is measured in terms of concrete actions taken by members of the couple in order to end their union. The total score is between 0 and 14. The higher the scores, the higher the risk of separation and marital distress. A threshold of 8 is considered to be a severe indicator of separation.
Change in Marital Status Inventory (MSI)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Partners
  The MSI is used to measure marital stability in a couple. It comprises a series of 14 items (with inverted items) in a "true" or "false" format thus aiming to assess the risk of separation in this couple (e.g., I very often have ideas of divorce, until once a week or more). Marital distress is measured in terms of concrete actions taken by members of the couple in order to end their union. The total score is between 0 and 14. The higher the scores, the higher the risk of separation and marital distress. A threshold of 8 is considered to be a severe indicator of separation.
Change in Dyadic Adjustment Scale (DAS-4)-Gambler | in the last seven days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  The Dyadic Adjustment Scale is an ultra-brief measure degree of marital satisfaction within the couple.
  The short version is made up of only 4 items (considered divorce, estimation of the quality of the relation, confide to mate, degree of happiness): three of which are on a 6-point Likert scale ranging from 0 (all the time) to 5 (never) , while the final item is on a 7-point scale ranging from 0 (extremely happy) to 6 (perfect).
  Theoretically possible maximum score of 21, and minimum 0. Scores lower than 11 indicating relationship distress, scores between 12 and 14 corresponding to medium satisfaction and scores upper 15 indicating good marital satisfaction.
Change in Dyadic Adjustment Scale (DAS-4)-Partner | in the last seven days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Partners
  The Dyadic Adjustment Scale is an ultra-brief measure degree of marital satisfaction within the couple.
  The short version is made up of only 4 items (considered divorce, estimation of the quality of the relation, confide to mate, degree of happiness): three of which are on a 6-point Likert scale ranging from 0 (all the time) to 5 (never) , while the final item is on a 7-point scale ranging from 0 (extremely happy) to 6 (perfect).
  Theoretically possible maximum score of 21, and minimum 0. Scores lower than 11 indicating relationship distress, scores between 12 and 14 corresponding to medium satisfaction and scores upper 15 indicating good marital satisfaction.
Change in Conjugal Support Questionnaire(CSQ)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  This questionnaire measures the quality of the support received and given perceived by the two members of the couple. It consists of a total of 8 questions, with a 5-point scale (1 = never; 5 = always). The total score shows support received and support gave. Higher is the result, more it indicates that the member of the couple gave support and receives it (score min = 0 and score max = 40).
Change in Conjugal Support Questionnaire(CSQ)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Partners
  This questionnaire measures the quality of the support received and given perceived by the two members of the couple. It consists of a total of 8 questions, with a 5-point Likert scale (1 = never; 5 = always). The total score shows support received and support gave. Higher is the result, more it indicates that the member of the couple gave support and receives it (score min = 0 and score max = 40).
Change in Gratitude Questionnaire (GQ-6)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  This questionnaire was modified to measure gratitude within the couple[1]. It has been adjusted to take into account gratitude towards partner instead of non-specific gratitude towards others (e.g. there is so much about my partner that I could be grateful). The 6 items are answered using a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree). The negative items are recoded and the compilation of the scores is made from their average. A higher average score indicates a higher degree of gratitude towards the partner (max=42, min=7).
Change in Gratitude Questionnaire (GQ-6)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Partners
  This questionnaire was modified to measure gratitude within the couple [1]. It has been adjusted to take into account gratitude towards partner instead of non-specific gratitude towards others (e.g. there is so much about my partner that I could be grateful). The 6 items are answered using a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree). The negative items are recoded and the compilation of the scores is made from their average. A higher average score indicates a higher degree of gratitude towards the partner (max=42, min=7).
Change in Generosity Scale-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  This tool, made up of 4 items, assesses the frequency of gestures and expressions of generosity between the members of the couple (taking small gestures that bring pleasure, expressing respect, showing affection, showing forgiveness). Participants are asked to rate how often they engage in this type of behavior using a scale from 1 (always) to 5 (never). The scores are then reversed, indicating that a higher score suggests the presence of greater generosity of the member of the couple towards their partner(max=20, min=4).
Change in Generosity Scale-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Partners
  This tool, made up of 4 items, assesses the frequency of gestures and expressions of generosity between the members of the couple (taking small gestures that bring pleasure, expressing respect, showing affection, showing forgiveness). Participants are asked to rate how often they engage in this type of behavior using a scale from 1 (always) to 5 (never). The scores are then reversed, indicating that a higher score suggests the presence of greater generosity of the member of the couple towards their partner (max=20, min=4).
Change in World Health Organisation-Five Well-Being Index (WHO-5)-Gambler | in the last seven days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  The WHO-5 is a self-answered questionnaire that measures the general state of a person's mental health using 5 items. The raw score (0-25) is multiplied by four to get a final score where 0 represents the worst state of mental health and 100 the best.
Change in World Health Organisation-Five Well-Being Index (WHO-5)-Partner | in the last seven days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Partners
  The WHO-5 is a self-answered questionnaire that measures the general state of a person's mental health using 5 items. The raw score (0-25) is multiplied by four to get a final score where 0 represents the worst state of mental health and 100 the best.
Change in Psychological Distress Index from the Quebec Health Survey-Gambler | in the last seven days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  This instrument is used to measure psychological distress, including symptoms of depression and anxiety. For the purpose of the study, the 14-items version will be used. The respondent should answer based on their condition in the past seven days using a 3-point Likert-type scale ranging from 1 (never) to 3 (very often). The higher the score, the more it indicates the presence of psychological distress (max=42, min=14)
Change in Psychological Distress Index from the Quebec Health Survey-Partner | in the last seven days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Partners
  This instrument is used to measure psychological distress, including symptoms of depression and anxiety. For the purpose of the study, the 14-items version will be used. The respondent should answer based on their condition in the past seven days using a 3-point Likert-type scale ranging from 1 (never) to 3 (very often). The higher the score, the more it indicates the presence of psychological distress (max=42, min=14)
Change in Ways of Coping Questionnaire-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  This questionnaire aims to identify the coping strategies used to cope with gambling or substance use habits. The abridged version includes 21 items divided into three subscales: Social Support Seeking (6 items), Positive Reassessment / Problem Solving (9 items), and Distancing / Avoidance (6 items).All items are rated on a Likert-type scale from 0 to 3 (0 = not used; 3 = used a lot). A higher score on one of the scales indicates that the person tends to adopt the behavior described by the scale when trying to adapt to a stressful situation (max=63, min=0).
Change in Ways of Coping Questionnaire-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Partners
  This questionnaire aims to identify the coping strategies used to cope with gambling or substance use habits. The abridged version includes 21 items divided into three subscales: Social Support Seeking (6 items), Positive Reassessment / Problem Solving (9 items), and Distancing / Avoidance (6 items).All items are rated on a Likert-type scale from 0 to 3 (0 = not used; 3 = used a lot).A higher score on one of the scales indicates that the person tends to adopt the behavior described by the scale when trying to adapt to a stressful situation (max=63, min=0).
Change in History of Psychiatric Hospitalization-Gambler | in the last six months of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  This question (only one) is used to document the number of hospitalizations and use of psychiatric emergency services of the gambling spouse in the past six months.
Change in History of Psychiatric Hospitalization-Partner | in the last six months of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Partners
  This question (only one) is used to document the number of hospitalizations and use of psychiatric emergency services of the partner in the past six months.
Change in Judicial sphere-Gambler | in the last six months of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  This 8-item questionnaire makes it possible to document the legal history of the person (indictment, trial or sentence, incarceration) and, if necessary, the type of offense committed and the type of judicial measure (conditional release, probation, halfway house, etc.).
Change in Judicial sphere-Partner | in the last six months of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Partners
  This 8-item questionnaire makes it possible to document the legal history of the person (indictment, trial or sentence, incarceration) and, if necessary, the type of offense committed and the type of judicial measure (conditional release, probation, halfway house, etc.).
Change in History of addiction treatment-Gambler | in the last six months of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  The purpose of the 3 items in this questionnaire is to document the use of addiction services over the past six months.
Change in Empathic Concern subscale from the Interpersonal Reactivity Index (IRI-Short form)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  The IRI-short form is a self-reported tool aims to assess an individual's ability to empathize. The Empathic Concern subscale (4 items) is the affective dimension of empathy, it refers to the respondent's feelings of compassion and concern for others. Using a 5-point Likert scale ranging from 0 (Does not describe me well) to 4 (Describes me very well), participant rates how closely each statement matches their overall way of behaving. Some items are reversed-scored. Responses to each subscale are averaged to reveal aggregate scores for each subdimension, there is no overall score. A high score represents a high presentation of this characteristic in the participant (max=16, min=0).
Change in Empathic Concern subscale from the Interpersonal Reactivity Index (IRI-Short form)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Partners
  The IRI-short form is a self-reported tool aims to assess an individual's ability to empathize. The Empathic Concern subscale (4 items) is the affective dimension of empathy, it refers to the respondent's feelings of compassion and concern for others. Using a 5-point Likert scale ranging from 0 (Does not describe me well) to 4 (Describes me very well), participant rates how closely each statement matches their overall way of behaving. Some items are reversed-scored. Responses to each subscale are averaged to reveal aggregate scores for each subdimension, there is no overall score. A high score represents a high presentation of this characteristic in the participant (max=16, min=0).
Change in Alcohol, Smoking and Substance Involvement and Screening Test (ASSIST) of the World Health Organization (WHO)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  This 8-item tool is developed by a group of the World Health Organization (WHO) specialized in addiction. It detects the use of different substances from the partner and proposes a threshold above which reported consumption behaviors are problematic (low risk: 0-3 for drug use and 0-10 for alcohol use, moderate risk: between 4-26 for drug use and between 11-26 for alcohol use, high risk 27 and more for alcohol and drug use).
Change in Canadian Problem Gambling Severity Index (PGSI)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  The Canadian Problem Gambling Index (CPGI) is a 9-item measure with a 4-point Likert-type scale (0 = Never, 3 = Almost always). It asks questions about the partner's gambling habits in the last three months from four categories:
  Gambling involvement; Problem gambling behaviour; Adverse Consequences; Correlates of problem gambling.
  Scores for the nine items are summed, and the results are interpreted as follows: 0 = non-problem ; 1-4 = low risk; 5-7 = moderate risk; 8 and + (maximum 27) = probable pathological player.
Change in Strategies facilitating the cessation of gambling and/or substance use behaviors and strategies promoting gambling and/or substance use behaviors-Partners | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners This questionnaire was developped to better understand what strategies the partner has put in place in the last three months in an attempt to reduce the gambling/using behaviors of her spouse or the strategies that may promote gambling/using habits.
  Partners must answer a total of 76 items with a 11-point scale, "0" = "Never" or "Not at all" to "10" = "extremely" or "always".
  For strategies promoting gambling and/or substance use behaviors the scales are 1)minimizing gambling/using behaviors; 2)gambling/using with the gambler; 3)reinforcing the gambler following a win; 4)hiding gambling/using behaviours from others; 5)funding gambling/using behaviours ; 6)making gambling/using available to the gambler. For reinforcement of sober behaviors, the scales are: 1)punishing, insulting, or threatening; 2)asking to stop gambling/using; 3)reducing access and non-gambling/non-using activities; 4)valuing times when the gambler is not gambling.
Change in Attribution scale for my spouse's gambling and/or substance use behaviors-Partners | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  This 22-item questionnaire uses a 5-point Likert-type scale (1 = Totally disagree, 5 = Totally agree) to measure the attributions (how I explain my partner's gambling behaviors and relapses) of someone having a player as a spouse. For example, my partner went to play because he wants to make me angry. The higher the score, the more the partner explains his spouse gambling's behaviors in a way that is inappropriate (max=110). The lower the score, the more adequately the partner will be able to explain his spouse gambling's behaviors(min=22).
Change in Transgression-Related Interpersonal Motivations-18 (TRIM-18)-Partners | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  This questionnaire consists of 18 items that measure avoidance, revenge and kindness motivations to forgive a spouse who has committed a relational transgression. Partners are instructed to think about a hurtful transgression and then indicate their agreement with each item using a 5-point response option ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores in a scale indicate higher motivations in relation with transgression (revenge, avoidance or kindness; max=30, min=6).
Change in Level of trust in the partner | in the last seven days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  This item measures the level of trust a partner has in the spouse who is a gambler. The partner answers the following question : " In the last week, how much trust did you have in your partner ? ", with a 11-point scale ranging from 0 (not at all) to 10 (Extremely). A high score means high trust in the partner.
Change in Self-Forgiveness Dual-Process Scale-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  Self-forgiveness is one of the components of the forgiveness process within romantic relationships. This questionnaire is composed of 10 items with a 7-point scale (1 = strongly disagree and 7 = strongly agree). It is separated into two subscales, namely 1) the reorientation of my value and 2) the restoration of self-esteem. Higher score means higher self-forgiveness (max=70, min=10).
Change in The Brief Accessibility, Responsiveness and Engagement (BARE)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  This 12 items self-answered questionnaire measures attachment behaviors in the context of a love relationship. The respondent must evaluate his behavior as well as that of his/her partner. Behaviors that are measured include accessibility (physical and emotional availability), receptivity (attention and listening), and engagement (mutual unity and connection). A high score indicates secure attachment behaviors in the couple(max=60, min=12).
Change in Interaction about addiction-Gambler | in the last seven days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  This one item measures the extent to which the interactions with the spouse about addiction, in the last week, were constructive. It is answered on a 11-point scale ranging from 0 (not at all) to 10 (Extremely). A high score means a high level of constructive interactions.
Change in Communication about cravings and use behaviors of substances and/or gambling | in the last seven days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  This one item measures the extent to which a gambler have talked about his cravings or behaviors of use to his spouse in the last week. The item is answered on a 11-point scale ranging from 0 (not at all) to 10 (Extremely). A high score means a high level of communication about cravings and/or use behaviors.
Change in Communication Patterns Questionnaire (CPQ)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  The CPQ is a 35-item self-report measure in which couple members independently report their typical interaction patterns. The measure assesses interactions across three time periods : 1) when a problem arises, 2) during discussion of the problem and 3) after the discussion of the problem. It uses a 9-point Likert scale to indicate the likelihood of that particular pattern occuring.
  The items of the CPQ are most commonly used to generate four subscales : Constructive Communication (seven items), Mutual Avoidance (three items), and two demand/withdraw scales (Self-Demand/Partner Withdraw and Partner-Demand/ Self-Withdraw; three items each). A high score indicates more use of that communication pattern during conflict.
Change in Couples Communication Satisfaction Scale (CCSS)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  The CCSS is used to assess the satisfaction of both members of the couple with respect to communication processes and behaviors. It is made up of 12 items which are answered on a 5-point Likert-type scale (1 = not at all satisfied to 5 = extremely satisfied). The items generates five subscales : personal communication, self-emotional experience, my partner's contribution, my partner's responsiveness and communication characteristics. The total score can range from 12 to 60, a high score means a high level of satisfaction with the communication processes and behaviors in the couple.
Change in Marital Problem Solving Scale (MPSS)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  The MPSS has 9 items, which are answered on a 7-point scale. It is use to better understand the negotiation and conflict resolution skills that the couple members have used within their marital relationship in the last three months. The score varies between 9 and 63. A high score indicates a greater degree of perceived problem-solving skill within the marital relationship.
Change in Substance Use Recovery Evaluator (SURE)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  The SURE is a self-answered questionnaire that measures recovery from addiction in the last week and provide information on what is important to someone in recovery. In the context of the study, only the Self-care subscale. The 5-items are answered from 1 = 'A little of the time' or 'None of the time', 2 = 'A fair amount of the time', 3 = 'All of the time' or 'Most of the time', meaning it can result in a 5-15 score range. Higher score means higher self-care habits.
Change in World Health Organization Quality of Life Assessment Brief (WHOQOL)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  The brief version of the WHOQOL is a 24-item questionnaire that assesses quality of life across four dimensions : social relationships, environment, physical and psychosocial. The four domain scores denote an individual's perception of quality of life in each particular domain : the mean score of items within each domain is used to calculate the domain score. Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life).
Change in Snyder's State Hope Scale (SHS)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  The SHS is utilized to measure participants' current state of hope. It is a brief 6-item measure. Responses are rated on an 8-point ranging from 1 (definitely True) to 8 (definitely False) with higher scores indicative of greater state hopefulness(max=48, min=6).
Change in Social Provisions Scale (SPS-10)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  The SPS-10 is a 10-item questionnaire that is use to measure social support. Specifically, it assesses five forms of social provisions: attachment, guidance, social integration, reliable alliance and reassurance of worth. Each item is rated on a four-point Likert scale (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree). A continuous scale score is computed by summing responses to the 10 questions, with values ranging from 10 to 40. Higher scores can be interpreted as having higher levels of social support.
Change in Social Provisions Scale (SPS-10)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  The SPS-10 is a 10-item questionnaire that is use to measure social support. Specifically, it assesses five forms of social provisions: attachment, guidance, social integration, reliable alliance and reassurance of worth. Each item is rated on a four-point Likert scale (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree). A continuous scale score is computed by summing responses to the 10 questions, with values ranging from 10 to 40. Higher scores can be interpreted as having higher levels of social support.
Change in World Health Organization Quality of Life Assessment Brief (WHOQOL)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  The brief version of the WHOQOL is a 24-item questionnaire that assesses quality of life across four dimensions : social relationships, environment, physical and psychosocial. The four domain scores denote an individual's perception of quality of life in each particular domain : the mean score of items within each domain is used to calculate the domain score. Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life).
Change in Scale of perception of gambling and/or substance use and involvement for those around them-for Partners | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  This 12-item questionnaire is used to better understand how the partner explains 1) his partner's recovery (eg, gambling is like an illness, he always remains vulnerable), 2) his understanding of relapses (eg, throughout his life, he will always be at risk of having a gambling fall) as well as 3) his supporting role (eg, I must not help him manage his finances). It uses a 5-point Likert-type scale (1 = totally disagree and 5 = totally agree) and has reversed-score items. The higher the score, the more the partner has a more negative view of their spouse's recovery and of their involvement with them(max=60, min=12).
Change in Barriers to Forgiveness Scale (BFS)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  The BFS is a 20-item questionnaire that is designed to identify the reasons why it is difficult for a partner to forgive. It theorized that people do not forgive for both reactive reasons (the offence is too hurtful and morally repugnant) and active reasons (deliberately refusing to forgive to protect the self from power and identity threats). It uses a 5-point Likert-type scale (1 = strongly disagree and 5 = strongly agree). The higher the score, the greater the barrier to forgiveness (max=100, min=20).
Change in State Shame and Guilt Scale (SSGS)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  The SSGS is a self-rating scale of in-the-moment (state) feelings of shame, and guilt experiences. It comprises of 8 items based on a Likert-type scale to 5 from 1 (disagree) to 5 (very agree) that explore state guilt and shame. The higher the score, the more shame and guilt the person feels (max=40, min=8).
Change in The Brief Accessibility, Responsiveness and Engagement (BARE)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  This 12 items self-answered questionnaire measures attachment behaviors in the context of a love relationship. The respondent must evaluate his behavior as well as that of his/her partner. Behaviors that are measured include accessibility (physical and emotional availability), receptivity (attention and listening), and engagement (mutual unity and connection). A high score indicates secure attachment behaviors in the couple(max=60, min=12).
Change in Couples Communication Satisfaction Scale (CCSS)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  The CCSS is used to assess the satisfaction of both members of the couple with respect to communication processes and behaviors. It is made up of 12 items which are answered on a 5-point Likert-type scale (1 = not at all satisfied to 5 = extremely satisfied). The items generates five subscales : personal communication, self-emotional experience, my partner's contribution, my partner's responsiveness and communication characteristics. The total score can range from 12 to 60, a high score means a high level of satisfaction with the communication processes and behaviors in the couple.
Change in Self-care questionnaire (Tremblay, 2022)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  13 items measure self-care behaviors in the last week. The items are answered from 1 = 'A little of the time' or 'None of the time', 2 = 'A fair amount of the time', 3 = 'All of the time' or 'Most of the time', meaning it can result in a 5-15 score range. Higher score means higher self-care habits.
Change in Self-care questionnaire (Tremblay, 2022)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  13 items measure self-care behaviors in the last week. The items are answered from 1 = 'A little of the time' or 'None of the time', 2 = 'A fair amount of the time', 3 = 'All of the time' or 'Most of the time', meaning it can result in a 5-15 score range. Higher score means higher self-care habits.
Change in Marital Problem Solving Scale (MPSS)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  The MPSS has 9 items, which are answered on a 7-point Likert-type scale. It is use to better understand the negotiation and conflict resolution skills that the couple members have used within their marital relationship in the last three months. The score varies between 9 and 63. A high score indicates a greater degree of perceived problem-solving skill within the marital relationship.
Change in Communication Patterns Questionnaire (CPQ)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  The CPQ is a 35-item self-report measure in which couple members independently report their typical interaction patterns. The measure assesses interactions across three time periods : 1) when a problem arises, 2) during discussion of the problem and 3) after the discussion of the problem. It uses a 9-point Likert scale to indicate the likelihood of that particular pattern occuring.
  The items of the CPQ are most commonly used to generate four subscales : Constructive Communication (seven items), Mutual Avoidance (three items), and two demand/withdraw scales (Self-Demand/Partner Withdraw and Partner-Demand/ Self-Withdraw; three items each). A high score indicates more use of that communication pattern during conflict.
Change in Interaction about addiction-Partner | in the last seven days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  This one item measures the extent to which the interactions with the spouse about addiction, in the last week, were constructive. It is answered on a 11-point scale ranging from 0 (not at all) to 10 (Extremely). A high score means a high level of constructive interactions.
Change in The Experience in Close Relationship Scale short-form (ECR-S)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  It is recognized that the attachment style of each member of the couple can influence the forgiveness process, which is why it is necessary to measure it. The short version of the ECR has 12 items with a 7-point Likert-type scale (1 = strongly disagree and 7 = strongly agree). Higher scores on the Anxiety and Avoidant subscales indicate higher levels of attachment anxiety and attachment avoidance, respectively.
Change in The Experience in Close Relationship Scale short-form (ECR-S)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  It is recognized that the attachment style of each member of the couple can influence the forgiveness process, which is why it is necessary to measure it. The short version of the ECR has 12 items with a 7-point Likert-type scale (1 = strongly disagree and 7 = strongly agree). Higher scores on the Anxiety and Avoidant subscales indicate higher levels of attachment anxiety and attachment avoidance, respectively.
Change in Dyadic Trust Scale (DTS)-Partner | in the last seven days prior to admission, 6, 12 and 18 post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  The DTS is use to measure the level of trust within the couple. It is made up of 8 items (including 5 reversed items) with a 5-point Likert-type scale (1 = not applicable at all to 5 = fully). Higher score means higher trust within the couple (max=40, min=8).
Change in Dyadic Trust Scale (DTS)-Gambler | in the last seven days prior to admission, 6, 12 and 18 post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gambler
  The DTS is use to measure the level of trust within the couple. It is made up of 8 items (including 5 reversed items) with a 5-point Likert-type scale (1 = not applicable at all to 5 = fully). Higher score means higher trust within the couple (max=40, min=8).
Change in Conflict Tactics Scale-2 _ Physical Violence Issued by the spouse-Gamblers | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Gamblers
  The physical violence suffered is a subscale of the CTS-2 questionnaire which aims to assess the manifestations of physical violence committed against the Gambler in the last 3 months. It is made up of 18 items that are rated on a 7-point Likert scale (never happened = 0, 1 time = 1, 2 times = 2, 3 to 5 times = 3, 6 to 10 times = 4, 11 to 20 = 5, more than 20 times = 6). The total score corresponds to the average obtained on the 18 items, the higher it is, more it indicates that the respondent has suffered episodes of violence.
Change in Conflict Tactics Scale-2 _ Physical Violence Issued by the spouse-Partners | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for the Partners
  The physical violence suffered is a subscale of the CTS-2 questionnaire which aims to assess the manifestations of physical violence committed against the partner in the last 3 months. It is made up of 18 items that are rated on a 7-point Likert scale (never happened = 0, 1 time = 1, 2 times = 2, 3 to 5 times = 3, 6 to 10 times = 4, 11 to 20 = 5, more than 20 times = 6). The total score corresponds to the average obtained on the 18 items, the higher it is, more it indicates that the respondent has suffered episodes of violence.
Change in Perspective Taking subscale from the Interpersonal Reactivity Index (IRI-Short form)-Gambler | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Gamblers
  The IRI-short form is a self-reported tool aims to assess an individual's ability to empathize. The Perspective Taking subscale (4 items), the tendency to spontaneously adopt the psychological point of view of others, concerns its cognitive dimension. Using a 5-point Likert scale ranging from 0 (Does not describe me well) to 4 (Describes me very well), participant rates how closely each statement matches their overall way of behaving. Some items are reversed-scored. Responses to each subscale are averaged to reveal aggregate scores for each subdimension, there is no overall score. A high score represents a high presentation of this characteristic in the participant (max=16, min=0).
Change in Perspective Taking subscale from the Interpersonal Reactivity Index (IRI-Short form)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome Measure for Partners
  The IRI-short form is a self-reported tool aims to assess an individual's ability to empathize. The Perspective Taking subscale (4 items), the tendency to spontaneously adopt the psychological point of view of others, concerns its cognitive dimension. Using a 5-point Likert scale ranging from 0 (Does not describe me well) to 4 (Describes me very well), participant rates how closely each statement matches their overall way of behaving. Some items are reversed-scored. Responses to each subscale are averaged to reveal aggregate scores for each subdimension, there is no overall score. A high score represents a high presentation of this characteristic in the participant (max=16, min=0).
Change in Substance Use Recovery Evaluator (SURE)-Partner | in the last 90 days of admission, 6,12 and 18 months post-admission (The first admission is anticipated for april 2023 and the last in march 2024)
  Outcome measure for Partners
  The SURE is a self-answered questionnaire that measures recovery from addiction in the last week and provide information on what is important to someone in recovery. In the context of the study, only the Self-care subscale. The 5-items are answered from 1 = 'A little of the time' or 'None of the time', 2 = 'A fair amount of the time', 3 = 'All of the time' or 'Most of the time', meaning it can result in a 5-15 score range. Higher score means higher self-care habits.

CONTACTS AND LOCATIONS:
Overall Officials: Joël Tremblay, PhD, Principal Investigator — Université du Québec à Trois-Rivières
Locations (7):
- Canada (7):
  - Centre Intégré de Santé et de Services Sociaux de Lanaudière, Joliette, Quebec
  - Centre intégré de Santé et de Services Sociaux de Chaudière-Appalaches (CISSS-CA), Lévis, Quebec
  - Centre Universitaire Intégré de Santé et de Services Sociaux du Centre Sud de l'Ile de Montréal, Montreal, Quebec
  - Centre Intégré de Santé et de Services Sociaux de la Montérégie-Ouest, Saint-Hubert, Quebec
  - Centre Intégré de Santé et de Services Sociaux des Laurentides, Saint-Jérôme, Quebec
  - Centre Universitaire Intégré de Santé et de Services Sociaux de l'Estrie, Sherbrooke, Quebec
  - Centre Universitaire Intégré de Santé et de Services Sociaux de la Capitale Nationale, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mccullough ME, Emmons RA, Tsang JA. The grateful disposition: a conceptual and empirical topography. J Pers Soc Psychol. 2002 Jan;82(1):112-27. doi: 10.1037//0022-3514.82.1.112. PMID 11811629

DOCUMENTS (3):
  • Study Protocol (2024-04-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT05833503/Prot_005.pdf
  • Statistical Analysis Plan (2024-04-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT05833503/SAP_006.pdf
  • Informed Consent Form (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT05833503/ICF_007.pdf